CLINICAL TRIAL: NCT00978393
Title: A Randomised, Placebo-controlled, Double-blind, Incomplete Cross-over Design Trial to Evaluate the Effects of Liraglutide on Gastric Emptying, Energy Expenditure and Appetite, and to Evaluate Liraglutide Pharmacokinetics in Non-diabetic Obese Subjects
Brief Title: A Trial to Assess the Effect of Liraglutide on Gastric Emptying in Healthy Obese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-3630; 2008-003228-44 (EudraCT Number); U1111-1111-9119 (Other: WHO)
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Experimental)
  Interventions: Drug: liraglutide
- B (Experimental)
  Interventions: Drug: liraglutide
- C (Experimental)
  Interventions: Drug: liraglutide
- D (Experimental)
  Interventions: Drug: liraglutide
- E (Experimental)
  Interventions: Drug: liraglutide
- F (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — High dose liraglutide treatment (3.0 mg) followed by low dose liraglutide treatment (1.8 mg). Injected s.c. (under the skin) once daily in the evening.
  Arms: A
Drug: liraglutide — Low dose liraglutide treatment (1.8 mg) followed by high dose liraglutide treatment (3.0 mg). Injected s.c. (under the skin) once daily in the evening.
  Arms: B
Drug: liraglutide — Low dose liraglutide treatment (1.8 mg) followed by high placebo treatment (3.0 mg). Injected s.c. (under the skin) once daily in the evening.
  Arms: C
Drug: liraglutide — High placebo treatment (3.0 mg) followed by low dose liraglutide treatment (1.8 mg). Injected s.c. (under the skin) once daily in the evening.
  Arms: D
Drug: liraglutide — High dose liraglutide treatment (3.0) followed by low placebo treatment (1.8 mg). Injected s.c. (under the skin) once daily in the evening.
  Arms: E
Drug: liraglutide — Low placebo treatment (1.8 mg) followed by high dose liraglutide treatment (3.0 mg). Injected s.c. (under the skin) once daily in the evening.
  Arms: F

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the effect of liraglutide on gastric emptying, energy expenditure and appetite, and to evaluate liraglutide pharmacokinetics in non-diabetic obese volunteers. The trial is designed as a two-period, six-sequenced, crossover trial where the trial participant will enter two treatment periods with a wash-out period of 6-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 30.0-40.0 kg/m2
* Stable body weight (below 5 kg body weight change during past 3 month)
* Fasting plasma glucose below 7.0 mmol/L

Exclusion Criteria:

* Presence or history of cancer or any clinically significant cardiac, metabolic, renal, gastrointestinal, hepatic, endocrine, dermatological, haematological, or psychiatric diseases or disorders, considered by the Investigator to have influence of the results of this trial
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Current or history of treatment with medications that may cause significant weight gain, within 12 months prior to screening
* Use of weight lowering pharmacotherapy within the last 3 months prior to trial start
* Previous or scheduled (during the trial period) surgical treatment for obesity
* Diagnosed type 1 or type 2 diabetes
* Smoking habitually as judged by the Investigator
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods if not sterile or post-menopausal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-09-16 (Actual); Primary Completion 2011-06-08 (Actual); Study Completion 2011-06-08 (Actual)

PRIMARY OUTCOMES:
Gastric emptying measured as AUC0-300min of paracetamol postprandial concentration profiles during a standardised meal test with intake of 1.5 g paracetamol | after 35 days of treatment

SECONDARY OUTCOMES:
Gastric emptying: Cmax and AUC0-60min/AUC0-300min of paracetamol postprandial concentration profiles | after 35 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Maastricht, Netherlands

REFERENCES:
- [Result] van Can J, Sloth B, Jensen CB, Flint A, Blaak EE, Saris WH. Effects of the once-daily GLP-1 analog liraglutide on gastric emptying, glycemic parameters, appetite and energy metabolism in obese, non-diabetic adults. Int J Obes (Lond). 2014 Jun;38(6):784-93. doi: 10.1038/ijo.2013.162. Epub 2013 Sep 3. PMID 23999198
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com